CLINICAL TRIAL: NCT02481284
Title: Microcirculatory Evaluation of the Abdominal Skin in Breast Reconstruction With Deep Inferior Epigastric Artery Perforator Flap
Brief Title: Microcirculation of the Abdominal Skin After Deep Inferior Epigastric Artery Perforator Flap Procedure
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kim Alexander Tønseth, Head of Department, Oslo University Hospital
Other Study IDs: CAIngvaldsen
Record Dates: First submitted 2015-05-11; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Breast Reconstruction; Skin Perfusion
Keywords: Breast reconstruction; Deep inferior epigastric artery perforator flap; Skin perfusion; Plastic and reconstructive surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laser Doppler Perfusion Imaging: 20 consequetive cases undergoing breast reconstruction with Deep inferior epigastric artery perforator flap who had evaluation of the microcirculation of the abdominal skin with laser Doppler perfusion imaging
  Interventions: Device: Laser Doppler perfusion imaging

INTERVENTIONS:
Device: Laser Doppler perfusion imaging — LDPI is an extension of laser Doppler flowmetry (LDF) and was developed to generate a colour-coded perfusion image in a large area of skin.

SUMMARY:
The purpose of this study was to perform a quantitative perfusion study of the undermined abdominal skin in deep inferior epigastric artery perforator flap breast reconstruction patients in order to obtain more knowledge on perfusion dynamics. Laser Doppler perfusion imaging (LDPI) was used to evaluate this.

Microcirculatory changes were monitored in the abdominal skin of 20 consecutive patients. Measurements were taken and recorded within four standardized zones covering the skin between the xiphoid process and the upper incisional boundary of the flap (zone 1-4; cranial to caudal).

DETAILED DESCRIPTION:
Background: No studies have assessed the perfusion of the undermined abdominal skin in breast reconstruction with deep inferior epigastric artery perforator flap. A greater understanding of the procedure's impact on the perfusion of the abdominal skin can be valuable in predicting areas susceptible to necrosis.

Methods: Microcirculatory changes were monitored in the abdominal skin of 20 consecutive patients undergoing breast reconstruction with a deep inferior epigastric artery perforator flap. Quantitative mapping was performed with laser Doppler perfusion imaging at seven set intervals. Measurements were taken and recorded within four standardized zones covering the skin between the xiphoid process and the upper incisional boundary of the flap (zone 1-4; cranial to caudal).

ELIGIBILITY:
Inclusion Criteria:

* Secondary, unilateral breast reconstruction with a DIEAP
* All smokers stopped smoking 4 weeks prior to surgery

Exclusion Criteria:

* Metastatic disease
* Bilateral breast reconstruction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 20 women consecutively undergoing secondary, unilateral breast reconstruction with a DIEAP flap were identified and recruited to participate in the study. The patients were informed about of risks and benefits and gave written consent prior to participation. All smokers stopped smoking 4 weeks prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Perfusion of the abdominal zones measured in mean perfusion units | Preoperative
Perfusion of the abdominal zones measured in mean perfusion units | two hours (After raising the flap)
Perfusion of the abdominal zones measured in mean perfusion units | Three hours (After undermining)
Perfusion of the abdominal zones measured in mean perfusion units | Five hours (After abdominal closure)
Perfusion of the abdominal zones measured in mean perfusion units | Postoperative day 1 (POD1)
Perfusion of the abdominal zones measured in mean perfusion units | Postoperative day 3 (POD3)
Perfusion of the abdominal zones measured in mean perfusion units | Postoperative day 7 (POD7)

CONTACTS AND LOCATIONS:
Overall Officials: Kim A Tønseth, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Department of Plastic and Reconstructive Surgery, Oslo, Oslo County, Norway